# **Cover page**

# Title:

Associations between time to reduction and complications in patients with dislocated total hip arthroplasty: A protocol for an observational cohort study

# **NCT** number:

Not available

# Date:

4th March 2025

# Associations between time to reduction and complications in patients with dislocated total hip arthroplasty:

A protocol for an observational cohort study

Rikke Helene Frølund. Bjulf<sup>1</sup>, Rasmus Linnebjerg. Knudsen<sup>1</sup>, Aurelien Xuan Rosendal. Bahuet<sup>1</sup>, Mathias Therkel Steensbæk<sup>1</sup>, Anne-Sofie Linde Jellestad<sup>1</sup>, Tazio Maleitzke<sup>3</sup>, Kai Henrik Wiborg Lange<sup>1,2</sup>, Markus Harboe Olsen<sup>4,5</sup>, Anders Peder Højer Karlsen<sup>2,6</sup> Lars Hyldborg Lundstrøm<sup>1,2</sup>, Anders Kehlet Nørskov<sup>1,2</sup>

Correspondence: Rikke Helene Frølund Bjulf, Department of Anesthesiology, Copenhagen University Hospital – North Zealand, Hillerød, Dyrehavevej 29, 3400 Hillerød, Denmark. Email: rikke.helene.froelund.bjulf.01@regionh.dk

<sup>&</sup>lt;sup>1</sup>Department of Anesthesiology, Copenhagen University Hospital – North Zealand, Hillerød, Denmark

<sup>&</sup>lt;sup>2</sup>Department of Clinical Medicine, University of Copenhagen, Copenhagen, Denmark

<sup>&</sup>lt;sup>3</sup> Department of Orthopaedic Surgery Copenhagen University Hospital Hvidovre University of Copenhagen

<sup>&</sup>lt;sup>4</sup>Department of Neuroanaesthesiology, The Neuroscience Centre, Copenhagen University Hospital-Rigshospitalet, Denmark

<sup>&</sup>lt;sup>5</sup>Copenhagen Trial Unit, Centre for Clinical Intervention Research, The Capital Region, Copenhagen University Hospital - Rigshospitalet, Copenhagen, Denmark

<sup>&</sup>lt;sup>6</sup>Department of Anesthesiology and Intensive Care Medicine, Copenhagen University Hospital- Bispebjerg, Denmark

# Table of contents

| Background | 4 |
|----------------------------|----|
| Objective | 5 |
| Methods | 5 |
| Study design | 5 |
| Setting and Population | 5 |
| Inclusions Criteria | 6 |
| Exclusion Criteria | 6 |
| Exposure and Outcomes | 6 |
| Exposure variables | 6 |
| Outcome measures | 6 |
| Variables | 7 |
| Data collection | 7 |
| Data handling | 7 |
| Statistical Analysis | 8 |
| Strengths and limitations | 9 |
| Publications | 9 |
| References | 10 |
| Appendix | 11 |
| Annendiy 1: Variable table | 11 |

### **Background**

Total hip arthroplasty (THA) is one of the most performed surgical procedures worldwide, with well-established efficacy in relieving joint pain and enhancing patient mobility. <sup>1-4</sup> Between 1995 and 2023, around 241,000 primary THA's were recorded in Denmark, averaging over 8,000 procedures annually. <sup>3</sup> An increasing number of THAs are performed in Denmark, with, approximately 14,000 in 2023, caused by a growing elderly population. <sup>3,5,6</sup> In Denmark, the proportion of patients experiencing a dislocation of their primary THA is around 3%, and 23% of 1,400 THA revision surgeries performed in 2023 were due to dislocation. <sup>3,7</sup>

Dislocation of THA is painful and can result in neurovascular damage, making immediate reduction essential. Furthermore recurrent dislocations, can lead to a decrease in quality of life.<sup>8,9</sup> Patients are usually elderly and frail with multiple comorbidities, making them susceptible to perioperative complications. <sup>10</sup> Delirium is a common postoperative complication in elderly patients and can lead to increased length of stay, admission to Intensive care unit and incidence of other complications such as pneumonia and death.<sup>11-13</sup>

In Denmark, the standard treatment for dislocated THA is closed reduction, mostly performed in the operating theatre under general anesthesia and with potential additional use of a neuromuscular blocking agent. However, general anesthesia presents both logistical and clinical challenges. It requires the availability of an operating theatre and experienced personnel, consideration of fasting regimes, and carries an increased risk of cardiovascular and respiratory complications. Despite the widespread use of general anesthesia, there is currently a lack of consensus on how to provide anesthesia for patients with THA dislocations in Denmark.

Outside of Denmark, closed reduction of dislocated THA is increasingly being performed in the emergency department under sedation. <sup>9,16</sup> This strategy presents potential advantages of reducing time to reduction along with hospital costs and length of stay, while freeing up resources in operating theatres. <sup>17-21</sup> However, sedation may induce complications such as, respiratory depression, apnea, aspiration, and other adverse events, that can be safely avoided in an operating theatre using general anesthesia. <sup>16,22,23</sup>

It remains unclear whether time to reduction, type of anesthesia and strategy for airway management are associated with increased risks of postoperative complications after closed reduction of dislocated THA.

# **Objective**

The aim of the study is to investigate the impact of time to closed reduction on both patient related and organizational factors. These include, length of stay, hospitalization, admission to intensive care unit, rehospitalizations, delirium, all-cause mortality, infection requiring hospital contact, and cardiovascular complications. We also intend to investigate whether different anesthetic strategies and airway management are associated with different complication rates.

We hypothesize that longer waiting time until reduction increase the post procedure length of stay, readmissions, and risk of complications.

### Methods

This protocol is developed in accordance with the principles outlined in STROBE (Strengthening the Reporting of Observational Studies in Epidemiology).<sup>24</sup>

### Study design

We will conduct a retrospective cohort study based on prospectively collected clinical data on patients presenting with THA dislocations who were treated with closed reduction in an operating theatre.

### **Setting and Population**

The cohort contains all adults presenting with a dislocated THA, who underwent closed reduction in an operating theatre with anesthesiology being involved, in public hospitals in the Capital and Zealand Regions of Denmark.

The study population is extracted from a dataset retrieved from the Electronic Health Record (EHR) system 'Sundhedsplatformen' (Epic Systems Corporation, WI, USA) from 1 January 2017 to 31 December 2024, including granular data from approximately 1.1 million anesthetic procedures.

### **Inclusions Criteria**

Patients are eligible for inclusion if they are 18 years of age or above, presented in the emergency department with a dislocated THA, and underwent subsequent closed reduction in the operating theatre with the involvement of anesthesiology.

### **Exclusion Criteria**

Patients are excluded if they:

- Were primarily booked for open surgical reduction.
- Did not have a complete case log (i.e. time of admission; referral to the operation theatre; anesthesia induction; discharge, etc.) and we were unable to recreate the log using simple code rules.

### **Exposure and Outcomes**

### Exposure variables.

- Time in minutes from admission to closed reduction.
- Time of day
- Weekday vs. weekend
- Airway management
- Anesthesia method(s)
- Neuromuscular blocking agent (Yes/No)

### Outcome measures

### Primary outcome

- Post procedure length of stay in minutes from closed reduction until discharge from the hospital.

### Secondary outcomes

- All-cause mortality at 90 days. (Y/N)
- Post procedure admission to the intensive care unit within 30 days (Y/N)
- Readmissions to hospital within 30 days (Y/N)
- Diagnosis with delirium or administration of haloperidol, olanzapine, risperidone, or quetiapine (as a surrogate for new onset delirium) (Y/N)

- Serum creatinine increase of more than 25 μmol/L within a period of less than 48 hours (as a surrogate for acute kidney failure) (Y/N)
- Infection requiring hospital contact.
- Cardiovascular complications (diagnosed arrythmia, myocardial infarction, cerebral ischemia or hemorrhage, pulmonary embolism or deep venous thrombosis)

### Variables

Patient demographics like age, sex, weight, height, BMI, American Society of Anesthesiology (ASA) classification, location (hospital), first-time dislocation/recurrent dislocation and comorbidity (diagnose codes at admission) will be retrieved for baseline statistics and adjustment in our multivariate statistical analyses.

A detailed list of variables is provided in **Appendix 1**.

### Data collection

The data is extracted from the EHR-system Sundhedsplatformen validated and cleaned. The patients are recorded when they are admitted to a public hospital in the Capital and Zealand Regions of Denmark, which contains one or more operations CSN-ID linked to an anesthesia CSN-ID (indicating that a procedure was performed with anesthesia).

The initial database extraction has been approved by 'Team for journaldata, videnskabsetik og forskningsstøtte, Region Hovedstaden' (Approval number R-23038250; 14 July 23). Furthermore, approval has been granted for the transfer of medical record data from the database to this research project (Approval number R-24079695; 13 December 24).

### Data handling

The dataset will undergo preprocessing and validation before analysis, including checks for missing values, duplicates, and errors. Only validated data will be used in the analysis to ensure accuracy and reliability.

Data will be stored in a secure database with restricted access. The dataset will be retained for a period and will be deleted once the study is completed.

### Statistical Analysis

Baseline data will be presented using descriptive statistics. For continuous variables, means and standard deviations (SDs) will be used to summarize data with normal distributions, and medians and interquartile range (IQR) for non-normally distributed data. Counts and percentages will represent categorical variables.

Linear regression models will be applied to assess the primary outcome of post procedure length of stay and other continuous outcomes.

Logistic regressions models with corresponding odds ratios (ORs) will be applied to assess the dichotomous secondary outcomes. To mitigate bias, we will adjust for relevant confounders in our statistical models and ensure data validation for the key variables, age, BMI, ASA-classification, comorbidities, site etc.

For all analyses we will present statistical tests as two-sided and consider a *p* value less than 0.05 statistically significant. For precision 95% confidence intervals will be presented.

For exposure variables with more than 10% missing data, multiple imputation will be employed to reduce potential bias. We will use baseline demographics (age, sex, BMI, ASA-classification, first-time dislocation/recurrent dislocation, site, and comorbidity) for imputation In cases where a patient undergoes multiple closed reductions during the observation period, we will conduct two analyses. The primary analysis will be based on each patient's first reduction event. A secondary analysis will utilize a linear mixed model for all reduction events regardless of multiple events by the same patient. In this latter analysis, patients will be included for each hospitalization that involves a dislocation requiring closed reduction.

In cases where missing data on outcome variables exceed 10%, we will impute worst-case and best-case scenarios and conduct sensitivity analyses to assess the impact of these imputations on our findings.

Statistical analyses will be performed using latest available stable version of R (R Core Team, Vienna, Austria).

## Strengths and limitations

This study offers several strengths. First, the retrospective design allows for a quick and cost-effective study, as data are already available. This allows for analysis of a large cohort of patients with dislocated THA and explores the impact of timing on outcomes such as length of stay, readmissions, and complications. Additionally, the use of an extensive patient database increases statistical power, enabling assessment of multiple outcomes across a broad sample.

Several limitations should be considered.

Selection bias may arise since the study relies on existing patient records potentially resulting in incomplete or non-representative data particularly for specific patient groups, e.g. those treated in emergency settings outside an operating theatre. This could limit the generalizability of the findings to a broader patient population.

Information bias may be present as clinical documentation might be inconsistent or incomplete, particularly regarding timing of reduction or complications. Additionally, patient identification relied on specific procedural codes for orthopedic surgery, which may have led to misclassification and potentially eligible patients being not correctly registered.

Confounding factors, such as comorbidities, may influence both the timing of reduction and clinical outcomes. Confounding by indication may occur if patients with more severe conditions are either delayed in receiving treatment or receive specific types of airway management, which may in turn affect both the timing of reduction and clinical outcomes. As an example, more frail or acute patients may experience shorter waiting times or specific airway interventions, while more healthy patients might face delays in treatment due to the less urgent nature of their condition. This could falsely appear to influence outcomes, when in fact, their poorer prognosis is due to their underlying condition rather than the treatment provided.

### **Publications**

Findings will be submitted for publication in an international, peer-reviewed journal relevant to the field of study.

### References

- 1. Stibolt, R.D., Jr., et al. Total hip arthroplasty for posttraumatic osteoarthritis following acetabular fracture: A systematic review of characteristics, outcomes, and complications. *Chin J Traumatol* **21**, 176-181 (2018).
- 2. Dainty, J.R., et al. Trajectories of pain and function in the first five years after total hip and knee arthroplasty: an analysis of patient reported outcome data from the National Joint Registry. Bone Joint J 103-b, 1111-1118 (2021).
- 3. (DHR), T.D.H.A.R. National Annual Report. (2023).
- 4. Price, A.J., et al. The use of patient-reported outcome measures to guide referral for hip and knee arthroplasty. *Bone Joint J* **102-b**, 941-949 (2020).
- 5. Kurtz, S., Ong, K., Lau, E., Mowat, F. & Halpern, M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. *J Bone Joint Surg Am* **89**, 780-785 (2007).
- 6. Rasmussen, M.B., El-Galaly, A., Daugberg, L., Nielsen, P.T. & Jakobsen, T. Projection of primary and revision hip arthroplasty surgery in Denmark from 2020 to 2050. *Acta Orthop* **93**, 849-853 (2022).
- 7. Kirurgi, D.O.S.D.S.f.H.-o.K. Total Hoftealloplastik, Referenceprogram (2006).
- 8. Kotwal, R.S., Ganapathi, M., John, A., Maheson, M. & Jones, S.A. Outcome of treatment for dislocation after primary total hip replacement. *The Journal of Bone & Joint Surgery British Volume* **91-B**, 321-326 (2009).
- 9. Germann, C.A., Geyer, D.A. & Perron, A.D. Closed reduction of prosthetic hip dislocation by emergency physicians. *Am J Emerg Med* **23**, 800-805 (2005).
- 10. Hopkins, T.J., et al. Associations between ASA Physical Status and postoperative mortality at 48 h: a contemporary dataset analysis compared to a historical cohort. *Perioper Med (Lond)* **5**, 29 (2016).
- 11. Inouye, S.K., Westendorp, R.G. & Saczynski, J.S. Delirium in elderly people. *Lancet* **383**, 911-922 (2014).
- 12. Schubert, M., et al. A hospital-wide evaluation of delirium prevalence and outcomes in acute care patients a cohort study. *BMC Health Serv Res* **18**, 550 (2018).
- 13. Inouye, S.K., et al. A multicomponent intervention to prevent delirium in hospitalized older patients. *N Engl J Med* **340**, 669-676 (1999).
- 14. Holler, C.P., Lohse, N. & Foss, N.B. Anaesthesia practice in Denmark for relocation of the dislocated hip after total hip arthroplasty. *Dan Med J* **65**(2018).
- 15. Harris, M. & Chung, F. Complications of general anesthesia. *Clin Plast Surg* **40**, 503-513 (2013).
- 16. Waseem, S., Ngu, A. & Patel, J. Emergency Department closed reduction of dislocated THR: the REDDTHR Prospective Multi-centre Study. *Hip Int* **34**, 633-640 (2024).
- 17. Dilbone, E.S., et al. Location of Initial Closed Reduction Attempt Significantly Increases Cost and Length of Stay in Total Hip Arthroplasty. *Arthroplast Today* **15**, 102-107 (2022).
- 18. Lawrey, E., Jones, P. & Mitchell, R. Prosthetic hip dislocations: is relocation in the emergency department by emergency medicine staff better? *Emerg Med Australas* **24**, 166-174 (2012).
- 19. Gagg, J., *et al.* Door to relocation time for dislocated hip prosthesis: multicentre comparison of emergency department procedural sedation versus theatre-based general anaesthesia. *Emerg Med J* **26**, 39-40 (2009).
- 20. Blokland, A., Van Den Akker, V., Van Der Poort, C., Somford, M. & Holkenborg, J. Results of Reduction of Dislocated Prosthetic Hips in the Emergency Department. *J Emerg Med* **62**, 462-467 (2022).
- 21. Sanchez-Sotelo, J., Haidukewych, G.J. & Boberg, C.J. Hospital cost of dislocation after primary total hip arthroplasty. *J Bone Joint Surg Am* **88**, 290-294 (2006).
- 22. Mathieu, N., et al. Is propofol a safe and effective sedative for relocating hip prostheses? *Emerg Med J* **26**, 37-38 (2009).

- 23. Saiz, A.M., Lum, Z.C. & Pereira, G.C. Etiology, Evaluation, and Management of Dislocation After Primary Total Hip Arthroplasty. *JBJS Rev* **7**, e7 (2019).
- von Elm, E., et al. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. *J Clin Epidemiol* **61**, 344-349 (2008).

# Appendix

# Appendix 1: Variable table

| Exposure variables | | | |
|---|---|---|---|
| Variable | Measurement | Definition | When |
| Time to reduction | Minutes, as a continuous | From arriving time in | From arriving time at the |
| | variable | the emergency | hospital until start of |
| | | department until the | procedure |
| | | start of procedure in | |
| | | the operating theater. | |
| Time of day | Nominal categorical | At arriving time at the | At arriving time at the |
| | variable, defined as 08- | hospital defined as | hospital |
| | 16, 16-00 or 00-08 | Day (08-16), evening | |
| | | (16-00) or nightshift | |
| | | (00-08) | |
| Weekday vs weekend | Nominal categorical | Defined as weekday | At arriving time at the |
| | variable | from Monday 08 to | hospital |
| | | Friday 00 and | |
| | | weekend Friday 00 to | |
| | | Monday 08. | |
| Airway management | Categorical variable, | The type of airway | At anesthesia induction |
| | defined as spontaneous | management | |
| | breathing, mask | categorized as | |
| | ventilation, elective | spontaneous | |
| | intubation, rapid | breathing, mask | |
| | sequence induction, or | ventilation, elective | |
| | laryngeal mask. | intubation, rapid | |

| | | sequence induction, or | |
|---|---|---|---|
| | | laryngeal mask. | |
| Anesthesia method(s) | Categorical variable, | Anesthesia method(s) | At anesthesia induction |
| | defined as propofol, | categorized as | |
| | etomidate, thiopental, | propofol, etomidate, | |
| | midazolam, ketamine, | thiopental, | |
| | sevoflurane, and | midazolam, ketamine, | |
| | desflurane. | sevoflurane, and | |
| | | desflurane. | |
| Neuromuscular blocking | Categorical variable | Neuromuscular | At anesthesia induction |
| agents | Rocuronium, | blocking agent | |
| | suxamethonium or non. | categorized as | |
| | | Rocuronium, | |
| | | suxamethonium or | |
| | | non. | |
| Primary outcomes | _ | | |
| Post-reduction length of stay | Minutes, as a continuous | Post procedure length | From procedure start until |
| | variable. | of stay. | hospital discharge up to 30 |
| | | | days after discharge. |
| Secondary outcomes | | | |
| All-cause mortality | Binary variable (Y/N) | 90 days all-cause | 90 days after closed |
| | | mortality | reduction |
| Admissions to Intensive care | Binary variable (Y/N) | Admissions to the | 30 days after the closed |
| unit | | intensive care unit | reduction |
| | | within 30 days after | |
| | | the closed reduction. | |
| Readmission | Binary variable (Y/N) | Readmission within | 30 days after discharge |
| | | 30 days after | |
| | | discharge | |
| Delirium | Binary variable (Y/N) | Defined as diagnose | Post procedure, during |
| | | of delirium (F05.x, | admission up to 30 day after |
| | | obtained from the | closed reduction. |

| | | diagnosis codes from | |
|---|---|---|---|
| | | the given admission) | |
| | | <b>or</b> the non-planned | |
| | | administration of | |
| | | haloperidol, | |
| | | olanzapine, | |
| | | risperidone, or | |
| | | quetiapine (as a | |
| | | surrogate for new | |
| | | onset delirium) | |
| Acute kidney failure | Binary variable (Y/N) | Defined as serum | Post procedure until 30 days |
| | | creatinine increase of | after discharge |
| | | more than 25 μmol/L | |
| | | within a period of less | |
| | | than 48 hours. or an | |
| | | increase in serum | |
| | | creatinine >1.5 times the | |
| | | baseline value, with | |
| | | baseline defined as the | |
| | | most recent | |
| | | measurement within the | |
| | | past 12 months (As a | |
| | | surrogate for acute | |
| | | kidney failure) | |
| Infection requiring hospital | Binary variable (Y/N) | Defined as diagnosed | Post procedure until 30 days |
| contact | | infection | after discharge |
| | | (postoperative | |
| | | infection (T81.4), | |
| | | pneumonia (J13.x- | |
| | | J18.x), Cystitis | |
| | | (N30.x, N39.0), sepsis | |

| | | (R65.x A40.x, A41.x), | |
|---|---|---|---|
| | | C. difficile (A04.7) | |
| | | obtained from the | |
| | | diagnose codes from | |
| | | the given admission) | |
| | | <b>or</b> administration of | |
| | | antibiotic treatment | |
| | | (as a surrogate for in- | |
| | | hospital infection | |
| Cardiovascular complications | Binary variable (Y/N) | Defined as diagnosed | From admission to 30 days |
| | | arrythmia (I47.x, | after discharge. |
| | | I48.x, I49.x), | |
| | | myocardial infarction | |
| | | (I21.x, I22.x), cerebral | |
| | | ischemia (I61.x, I63.x, | |
| | | I64.x), | |
| | | hemorrhage(T81), | |
| | | pulmonary | |
| | | embolism(I26.x) or | |
| | | deep venous | |
| | | thrombosis(I80.2) | |
| | | (obtained from the | |
| | | diagnosis codes from | |
| | | the given admission) | |
| Baseline variables | | | |
| Age | Years | | At admission |
| Sex | Male or female | | At admission |
| Weight | Kilograms | | At admission |
| Height | Centimeters | | At admission |
| BMI | Kg/m <sup>2</sup> | | At admission |
| ASA-score | ASA 1-6 | ASA I: Healthy | At admission |
| | | patient, ASA II: Mild | |

| | | systemic disease, ASA | |
|-------------|--------------------|------------------------|--------------|
| | | - | |
| | | III: Severe systemic | |
| | | disease, ASA IV: | |
| | | Severe systemic | |
| | | disease with constant | |
| | | threat to life, ASA V: | |
| | | Moribund patient, | |
| | | ASA VI: Declared | |
| | | brain-dead | |
| Comorbidity | Diagnosis codes at | Diagnose codes ad | At admission |
| | admission | admission | |
| | | (Hypertension (I10, | |
| | | I11. I12, I13, I14, | |
| | | I15), Osteoporosis | |
| | | (M80, M81, M82, | |
| | | M83), Diabetes (E10, | |
| | | E11, E12, E13, E14), | |
| | | Congestive Heart | |
| | | failure (I50.x), | |
| | | Ischaemic heart | |
| | | disease (I21.x, I22.x, | |
| | | I24.x, I25.x), | |
| | | Arrythmia (I47.x, | |
| | | I48.x I49.x), Chronic | |
| | | Obst. Pulm. Disease | |
| | | (J44), Cancer (C00- | |
| | | C97), Chronic kidney | |
| | | disease (N18), | |
| | | Cerebrovascular | |
| | | disease (I61.x, I63.x, | |
| | | I64.x), Mild liver | |
| | | disease (K70.x, K71.x, | |
| | 1 | <u> </u> | |

| | | K73.x, K74.x, K76.x), | |
|---|---|---|---|
| | | Moderate/severe liver | |
| | | disease (K72.x, I85.x), | |
| | | Alcohol-related | |
| | | disease (F10.x), Drug- | |
| | | related disease ( | |
| | | F11.x, F12.x, F13.x, | |
| | | F14.x, F16.x), | |
| | | Dementia (F00, F01, | |
| | | F02, F03), Parkinson | |
| | | disease (G20), | |
| | | Alzheimer (G30), | |
| | | Depression (F32.x- | |
| | | F33.x), Anxiety | |
| | | (F40.x-F41.x), | |
| | | Schizophrenia (F20.x) | |
| Location (Hospital) | OPIAD def. | Locations categorized | At admission. |
| | | in The Capital Region | |
| | | (Site A-F) and | |
| | | Zealand Region (Site | |
| | | G-I)of Denmark. | |
| First-time | Binary variable, First | | |
| dislocation/recurrent | time or recurrent | | |
| dislocation | dislocation. | | |